CLINICAL TRIAL: NCT03800095
Title: Early Palliative Care for Patients With Haematological Malignancies: A Randomised Prospective Study
Brief Title: Early Palliative Care for Patients With Haematological Malignancies
Acronym: CALVI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation Apicil (Other); Association des foulées de la Haute Lozère (Unknown); Association CEMSBM (Unknown); Connaître et Combattre les Myélodysplasies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-406; 2017-A02515-48 (Other: 2017-A02515-48)
Record Dates: First submitted 2018-09-13; First posted 2019-01-11 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Diffuse Large B Cell Lymphoma; Palliative Care
Keywords: Supportive care; Early palliative care; Quality of life; Symptoms management; Haematological malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional haematological care (Experimental): Patients with haematological malignancy Conventional haematological care
  Interventions: Drug: Early palliative care integration
- Conventional care associated with a monthly consultation (Experimental): Patients with haematological malignancy Conventional care associated with a monthly consultation realized by a palliative and supportive care team
  Interventions: Drug: Early palliative care integration

INTERVENTIONS:
Drug: Early palliative care integration — The follow-up time for each patient is 12 months with evaluation of the main objective by a standardized questionnaire: The Functional Assessment of Cancer Therapy-Anaemia (FACT-An) Scale at 6 months. Throughout the study, patients included will receive conventional haematological care and the interventional arm will benefit in addition to a monthly consultation by a palliative care team.

SUMMARY:
Patients suffering from haematological disease present symptoms of discomfort and currently benefit from palliative care skills only for the management of their end-of-life. However, in medical oncology, more and more studies tend to demonstrate the benefit on the quality of life of an early collaboration between the two specialties.

Investigator did the hypothesis that early integration of palliative care with conventional haematological care could decrease discomfort symptoms and add a real benefit on the patients' quality of life .

DETAILED DESCRIPTION:
Patients suffering from haematological disease present symptoms of discomfort and currently benefit from palliative care skills only for the management of their end-of-life. However, in medical oncology, more and more studies tend to demonstrate the benefit on the quality of life of an early collaboration between the two specialties.

Investigator did the hypothesis that early integration of palliative care with conventional haematological care could decrease discomfort symptoms and add a real benefit on the patients' quality of life .

ELIGIBILITY:
Inclusion Criteria:

* Patients are over 70 years old
* Patients from being diagnosed with acute myeloid leukemia and high-risk myelodysplastic syndrome or after the third line of therapy for high-grade lymphoma.

Exclusion Criteria:

* All patients with a curative project (induction chemotherapy ou allogenic transplantation)
* All patients in a terminal palliative status
* Patients who don't speak French,
* Patients not able to read and write
* Patients who don't agree to participate in the protocol
* Patients with psychiatric troubles or cognitive disorders
* Patients under guardianship or curatorship, deprived of freedom or under justice protection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-08-14 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life evaluation: standardized questionnaire | at 6 months
  Evaluation of quality of life by a standardized questionnaire : Functional Assessment of Cancer Therapy-Anemia (FACT-An). The higher is the score the better is the quality of life. FACT-An is composed by five subscales: Physical Well-Being [score range 0-28], Social/Family Well-Being [score range 0-28], Emotional Well-Being [score range 0-24], and Functional Well-Being [score range 0-28] and specific questions concerning anemia [score range 0-80]. The score at each items is summed. The sum is multiplied par the number of items in the subscale and then divided by the number of items answered. This produces the subscale score. The subscale scores are added to derive total score [score range 0-188].

SECONDARY OUTCOMES:
Presence of discomfort symptoms | at Day 0, 3 months, 6 months, 9 months, 12 months
  evaluated by Edmonton scale (depressive syndrome measured by the geriatric depression scale GDS)
overall survival | at day 1 : from the randomization until the date of death or until 1 year [study end].
Satisfaction of the care pathwaydesired by the patient | at 12 months or death
  matching between patients desires writing in the medical file and the providing care
cost-effectiveness analysis | at 12 months or death
  The cost criteria selected will be all the direct medical costs inherent in care in both arms (costs of hospitalizations, consultations, treatments, medical devices).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CH Jacques Lacarin, Vichy